CLINICAL TRIAL: NCT03353675
Title: A Phase II Study Evaluating the Efficacy and the Safety of First-line Chemotherapy Combined With TG4010 and Nivolumab in Patients With Advanced Non-squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study Evaluating the Efficacy and the Safety of First-line Chemotherapy Combined With the Therapeutic Vaccine Named TG4010 and Nivolumab in Patients With Advanced Non-squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transgene (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG4010.24
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: Metastatic NSCLC; Advanced lung malignancy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TG4010; Drug Therapy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TG4010/Chemotherapy/Nivolumab (Experimental)
  Interventions: Biological: TG4010; Drug: Chemotherapy; Drug: Nivolumab

INTERVENTIONS:
Biological: TG4010 — 1 dose (1x1E+08) Subcutaneous injection/week over 6 weeks then 1 dose/3 weeks
Drug: Chemotherapy — Pemetrexed/Cisplatin or Carboplatin
  Pemetrexed maintenance
Drug: Nivolumab — 360 mg IV administration every 3 weeks

SUMMARY:
This is a multicenter, single arm, open label phase II study in treatment-naïve for advanced stage of the disease and immunotherapy-naïve patients with advanced non-squamous NSCLC and with < 50% of tumor cells expressing programmed death-ligand 1 (PD-L1) by immunohistochemical (IHC) staining.

ELIGIBILITY:
Principal Inclusion Criteria:

* Female or male patients age > 18 years-old
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1 at study entry
* Life expectancy of at least 3 months
* Histologically confirmed non-squamous NSCLC (adenocarcinoma, large cell carcinoma, undifferentiated carcinoma or other)
* Stage IIIB-IV cancer or delayed relapse of any stage not amenable to surgery or radiotherapy with curative intent.
* PD-L1 expression by immunohistochemistry in < 50% of tumor cells
* Patients must be chemotherapy-naïve for the advanced stage of the disease. Previous neoadjuvant and/or adjuvant chemotherapy is allowed for patients who successfully underwent complete radical surgery and if last treatment was administered more than 12 months prior to the start of the study treatment.
* At least one measurable lesion by CT scan based on RECIST 1.1 performed within 28 days prior to start of study treatment
* Adequate hematological, hepatic, and renal functions
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the start of study drug
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug plus 30 days for a total of 5 months posttreatment completion. Highly effective contraception are defined in the protocol.
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 90 days for a total of 7 months post-treatment completion

Principal Exclusion Criteria:

* Patients having central nervous system (CNS) metastases
* Patients with pericardial effusion
* Prior exposure to cancer immunotherapy including cancer vaccines, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-Lymphocyte antigen- 4 antibody or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways
* Patients with epidermal growth factor receptor (EGFR) activating mutations or anaplastic lymphoma kinase (ALK)- rearrangements leading to eligibility for tyrosine kinase inhibitor (TKI) treatment (tests mandatory)
* Prior history of other malignancy except basal cell carcinoma of the skin, cervical intra epithelial neoplasia, and other cancer curatively treated with no evidence of disease for at least 3 years
* Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of start of study treatment
* Patients with an active, known or suspected autoimmune disease
* Patient with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Patients with grade ≥ 2 neuropathy
* Signs or symptoms of infection within 14 days prior to start of study treatment or active infection requiring systemic therapy
* Positive serology for HIV or hepatitis C virus (HCV); presence in the serum of the antigens hepatitis B (HBs) at baseline
* Patient with any underlying medical condition that the treating physician considers might be aggravated by treatment or which is not controlled (e.g., elevated troponin or creatinine, uncontrolled diabetes)
* History of cardiovascular conditions within 12 months of enrollment
* Left ventricular ejection fraction less than the Lower Limit of Normal as assessed by echocardiography (or multigated acquisition (MUGA) scan)
* Patient with major surgery or radiotherapy within 3 weeks prior to the start of the study treatment. However, prior surgery or radiation therapy aimed at local palliation or attempted local disease control (except in case of thoracic radiotherapy) is permitted but has to be completed 2 weeks before treatment start
* Pregnant or nursing (lactating) women
* Patients with an organ allograft
* Any known allergy to eggs, gentamicin or history of allergy or hypersensitivity to study drug components
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Charlotte, Charlotte, North Carolina
  - Nashville, Nashville, Tennessee
- Libramont, Libramont, Belgium
- France (4):
  - Créteil, Créteil
  - Mulhouse, Mulhouse
  - Rennes, Rennes
  - Strasbourg, Strasbourg
- Hungary (2):
  - Budapest, Budapest
  - Szekesfehervar, Székesfehérvár

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 study sites in United States, 4 sites in France, 2 sites in Hungary and 1 site in Belgium.
Pre-assignment Details: A total of 44 participants were enrolled and treated with at least one administration of each study drug.
Groups:
- TG4010/Chemotherapy/Nivolumab: TG4010: 1 dose (1x1E+08) Subcutaneous injection/week over 6 weeks then 1 dose/3 weeks
  Chemotherapy: Pemetrexed/Cisplatin or Carboplatin
  Pemetrexed maintenance
  Nivolumab: 360 mg IV administration every 3 weeks
Period: Overall Study
Arm/Group | TG4010/Chemotherapy/Nivolumab
Started | 44
Completed | 40
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 6
  Hungary | 6
  United States | 6
  France | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — ECOG PS 0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  participants
    ECOG PS 0 | 21
    ECOG PS 1 | 23
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 24.4 [15 to 37]
PD-L1 percentage of stained cells [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay (method Dako PD-L1 IHC 22C3 pharmDx assay kit) using tumor tissue from an archival or newly obtained biopsy. Participants with PD-L1 expression ≤50% of tumor cells were eligible to the study.
  Participants
    <1 | 22
    1 - <50 | 22
    ≥50 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Percentage of participants whose best overall response is complete response or partial response using RECIST 1.1. confirmed by a second scan no less than 4 weeks after the criteria for response are first met.
  Complete response: disappearance of all lesions and no new lesions. Partial response: decrease of at least 30% in the sum of the diameters of measurable lesions taking as reference the baseline sum of diameters, no progression of non-measurable lesions and no new lesions.
Time Frame: 15 months
Population: The Evaluable Patient's Population is the primary population for efficacy analyses. Evaluable Patient's Population consists of all participants without major protocol deviation and have at least one baseline and one post-baseline evaluable CT-scan after study treatment start except early disease progression and death due to lung cancer.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 40
percentage of participants | 32.5 [20.4 to 46.6]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from the date of the first study drug administration to the date of first documented tumor progression or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  The Kaplan-Meier estimator was used to estimate median PFS and its confidence interval.
Time Frame: 28 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 40
Months | 5.7 [1.5 to 11.1]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants whose best overall response is either complete response, partial response or stable disease. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan or MRI: Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions and no measurable non-target lesions; Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD).
Time Frame: 15 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 40
percentage of participants | 75.0 [61.3 to 85.8]

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from the first study drug administration to the date of death due to any cause.
  The Kaplan-Meier estimator was used to estimate median OS and its confidence interval.
Time Frame: 28 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 40
Months | 14.9 [8.0 to NA] — The upper limit of 95% confidence interval for overall survival was not reached by the end of the study period because too few participants with events to calculate upper confidence interval.

5. Secondary Outcome: Duration of Overall Response (DoR)
Description: Time from first documented response (complete response or partial response) until documented disease progression or death due to lung cancer.
Time Frame: 28 months
Population: Responders: all evaluable participants with complete response or partial response. The start date was the date of first documented response (complete response or partial response) and the end date was the date of first documented disease progression. If no progression has been observed at the cut-off date of analysis or at the date when a subsequent cancer therapy was started, duration of response was censored at the date of the last evaluable tumor assessment.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 13
Weeks | 74.9 [19.4 to 92.6]

6. Secondary Outcome: Number of Participants With Adverse Events or Abnormalities
Description: The assessment of safety of the combination was based mainly on the frequency of adverse events, serious adverse events, adverse events of special interest (Injection site reaction, fatigue, pyrexia, infusion-related reactions and diarrhea), immune-mediated adverse events and laboratories abnormalities.
Time Frame: 28 months
Population: Safety population (all treated participants)
Measure: Count of Participants; unit: Participants
Arm/Group | TG4010/Chemotherapy/Nivolumab
Number analyzed (Participants) | 44
Participants
  Adverse events | 44
  Serious adverse events | 28
  Adverse events of special interest | 37
  Immune-mediated adverse events | 14
  Grade 3/4 laboratories abnormalities | 31

ADVERSE EVENTS:
Time Frame: Collection of adverse events / serious adverse events starts from the date of signature of the informed consent form up to the safety follow-up visits (100 days after the last administration of any study treatment administration). Timeframe was approximately 28 months.
Arm/Group | TG4010/Chemotherapy/Nivolumab
All-Cause Mortality (participants affected / at risk) | 28/44
Serious Adverse Events (participants affected / at risk) | 28/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG4010/Chemotherapy/Nivolumab (N=44)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
AUTOIMMUNE COLITIS (Gastrointestinal disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DUODENITIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 9 (9)
FATIGUE (General disorders) | 2 (2)
CONDITION AGGRAVATED (General disorders) | 1 (1)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
BARTHOLINITIS (Infections and infestations) | 1 (1)
BRAIN ABSCESS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG4010/Chemotherapy/Nivolumab (N=44)
ANAEMIA (Blood and lymphatic system disorders) | 24 (43)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 14 (21)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 13 (20)
HYPOTHYROIDISM (Endocrine disorders) | 4 (4)
LACRIMATION INCREASED (Eye disorders) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (5)
CONSTIPATION (Gastrointestinal disorders) | 16 (17)
DIARRHOEA (Gastrointestinal disorders) | 17 (23)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 26 (31)
STOMATITIS (Gastrointestinal disorders) | 7 (8)
VOMITING (Gastrointestinal disorders) | 8 (10)
ASTHENIA (General disorders) | 3 (3)
FATIGUE (General disorders) | 29 (39)
INJECTION SITE ERYTHEMA (General disorders) | 5 (6)
INJECTION SITE PAIN (General disorders) | 5 (5)
INJECTION SITE REACTION (General disorders) | 6 (6)
OEDEMA PERIPHERAL (General disorders) | 9 (11)
PYREXIA (General disorders) | 5 (7)
CONJUNCTIVITIS (Infections and infestations) | 5 (5)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5)
BLOOD CREATININE INCREASED (Investigations) | 7 (7)
LIPASE INCREASED (Investigations) | 3 (3)
WEIGHT DECREASED (Investigations) | 8 (8)
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 (15)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 (13)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
DIZZINESS (Nervous system disorders) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 8 (8)
HEADACHE (Nervous system disorders) | 9 (9)
PARAESTHESIA (Nervous system disorders) | 8 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (13)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (14)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (5)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 7 (7)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 7 (9)
FLUSHING (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT03353675/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT03353675/SAP_001.pdf